CLINICAL TRIAL: NCT02666417
Title: Testing Iron Absorption From a New Micronutrient Powder Containing Galacto-oligosaccharides (GOS) for Fortification of Infant Foods in Sub-Saharan Africa
Brief Title: Iron Absorption From a Micronutrient Powder Containing Galacto-oligosaccharides (GOS)
Acronym: FeGOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Jomo Kenyatta University of Agriculture and Technology (Other); International Centre for Behavioural Studies (Unknown); Msambweni District Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FeGOS_KP; NCT03357510 (obsolete NCT alias)
Record Dates: First submitted 2016-01-20; First posted 2016-01-28 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Anemia, Iron-Deficiency
Keywords: Iron fortification; Anemia; Iron Deficiency; Iron Absorption; Prebiotics; Stable isotopes
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia; Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MNP+iron and test meal (Active Comparator): The MNP contains 400 μg Vitamin A, 5 μgVitamin D, 5 mg Tocopherol Equivalent, 0.5 mg Thiamine, 0.5 mg Riboflavin, 0.5 mg Vitamin B6 , 90 μg Folic Acid,6 mg Niacin, 0.9 μg Vitamin B12, 30 mg Vitamin C, 0.56 mg Copper, 90 μg, Iodine, 17 μg Selenium, 4.1 mg Zinc, 190 Phytase-units, plus 2.5 mg Fe as FeFum and 2.5 mg Fe as NaFeEDTA, maltodextrin carrier (added up to 11g)
  Iron compound added to the test meal: Test meal A will contain 2.5 mg 57Fe as ferrous fumarate and 2.5 mg of iron as NaFeEDTA (given as 1.5 mg 56Fe and 1 mg 58Fe). Test meal B will contain 5 mg iron in form of FeSO₄ (3 mg 56Fe and 2 mg 54Fe).
  Interventions: Dietary Supplement: Fortified maize porridge (MNP+iron)
- MNP+iron+GOS and test meal (Active Comparator): The MNP contains 400 μg Vitamin A, 5 μgVitamin D, 5 mg Tocopherol Equivalent, 0.5 mg Thiamine, 0.5 mg Riboflavin, 0.5 mg Vitamin B6 , 90 μg Folic Acid,6 mg Niacin, 0.9 μg Vitamin B12, 30 mg Vitamin C, 0.56 mg Copper, 90 μg, Iodine, 17 μg Selenium, 4.1 mg Zinc, 190 Phytase-units, plus 2.5 mg Fe as ferrous fumarate and 2.5 mg Fe as NaFeEDTA, plus 7.5 g of galacto-oligosaccharides given as 10.5 g GOS-75, maltodextrin carrier (added up to 11g)
  Iron compound added to the test meal: Test meal A will contain 2.5 mg 57Fe as ferrous fumarate and 2.5 mg of iron as NaFeEDTA (given as 1.5 mg 56Fe and 1 mg 58Fe). Test meal B will contain 5 mg iron in form of FeSO₄ (3 mg 56Fe and 2 mg 54Fe).
  Interventions: Dietary Supplement: Fortified maize porridge (MNP+iron+GOS)

INTERVENTIONS:
Dietary Supplement: Fortified maize porridge (MNP+iron) — Maize porridge will be home-fortified with the MNP + iron. Maize porridge for the test meal will be fortified with labelled iron compounds
  Arms: MNP+iron and test meal
Dietary Supplement: Fortified maize porridge (MNP+iron+GOS) — Maize porridge will be home-fortified with the MNP + iron + GOS. Maize porridge for the test meal will be fortified with labelled iron compounds
  Arms: MNP+iron+GOS and test meal

SUMMARY:
Infants and young children in sub-Saharan Africa have high rates of iron deficiency anemia (IDA), which adversely affects their growth and cognitive development. In-home iron fortification of complementary foods using micronutrient powders (MNPs) reduces risk for IDA. However, in areas with a high burden of infectious diseases iron may increase the risk of unfavorable gut microbiota composition possibly influencing diarrhea prevalence. Thus, there is an urgent need to find safer formulations of iron fortification for African infants. The investigators recently finished a randomized, double blind controlled intervention trial in Kenya where the investigators tested whether the addition of galacto-oligosaccharides (GOS) in a MNP containing 5 mg of iron protects against the adverse effects of the iron on the infant gut microbiome and gut inflammation (ClincalTrails.gov Identifier: NCT02118402). Prebiotics are also potential enhancers of colonic iron absorption. Therefore, to complement the intervention study, the present study will compare iron absorption from the combination of sodium iron EDTA (NaFeEDTA) and ferrous fumarate (FeFum) with and without prior consumption GOS or 3 weeks. The investigators will enroll 80 Kenyan infants from Kwale County, aged 6-14 months of whom 40 infants will consume maize porridge blended with MNP containing iron and 40 infants will receive a porridge mixed with MNP containing iron+GOS. After 3 weeks of MNP consumption, two test meals will be fed on two consecutive mornings, and will consist of maize porridge containing isotopically labeled FeFum and NaFeEDTA or isotopically labeled ferrous sulfate (FeSO₄), respectively. Fourteen days after the second test meal administration, a whole blood sample will be collected by venipuncture for iron isotopic analysis. Iron and inflammation status parameter will be determined at baseline and endpoint. A stool sample will be collected at baseline and on the first test meal day. The gut microbiome, fecal pH and fecal SCFAs profile will be analyzed. Knowing the expected iron absorption from the iron and GOS containing MNP will inform decisions on type of iron compound and dosing regimens for MNPs to allow the lowest iron dose to be used but still cover the infant requirement for absorbed iron.

DETAILED DESCRIPTION:
Iron absorption from two iron-fortified maize-based test meals will be measured in two groups of 40 infants (total N=80). Infants will be recruited at Msambweni District Hospital and communities served by Msambweni District Hospital in southern coastal Kenya. In group 1, iron absorption is measured after 3 weeks of MNP consumption containing 5 mg iron in form of NaFeEDTA (2.5 g) and FeFum (2.5 g) but no GOS. In group 2, iron absorption is measured after 3 weeks of MNP consumption containing 5 mg iron in form of NaFeEDTA (2.5 g) and FeFum (2.5 g) and 7.5 g GOS. Iron absorption is measured as the incorporation of stable isotopes into erythrocytes at least 14 days after the test meal administration.

At baseline, a blood sample will be collected from potential study participants for the determination of the following iron and inflammation status parameters: hemoglobin (Hb), plasma ferritin (PF), soluble transferrin receptor (sTfR), zinc protoporphyrin (ZnPP), C-reactive protein (CRP), alpha-1-acid glycoprotein (AGP). Anthropometrics (height, weight, mid-upper arm and head circumference) will be measured, and demographics, the medical history and the feeding habits will be assessed using a questionnaire. On day 1, infants will be enrolled and randomized into the two groups, and then start the intervention. The infants will consume 1 MNP sachet added to maize porridge per day for a total of 5 weeks. A stool sample will be collected on day 1 for the determination of gut microbiota composition, fecal pH and fecal SCFAs. After 3 weeks of MNP consumption, the two isotopically labelled test meals will be fed to the infants by their caregivers under supervision of the research team on two consecutive mornings between 7 and 8 am. Test meal A will contain 2.5 mg 57Fe in form of FeFum and 2.5 mg iron as NaFeEDTA (given as 1.5 mg 56Fe and 1 mg 58Fe). Test meal B will contain 5 mg iron in form of FeSO₄ (3 mg of 56Fe and 2 mg of 54Fe). The test meals will consist of maize porridge (5-10% dry weight) and mineral water (30 ml) and will be randomly administered on the two consecutive days (AB or BA). Overnight, only breast milk will be allowed to the infant and no breast milk will be given at least 3 h before test meal administration. Infants will not be allowed to eat or drink for 2 h after the test meal. On the day of the first test meal, a stool sample will be collected and analyzed for gut microbiota composition, fecal pH and fecal SCFAs. Fourteen days after the second test meal administration, 3 ml of whole blood will be collected by venipuncture for iron isotopic analysis and iron and inflammation status. Anthropometrics and the baseline questionnaire will be repeated. Compliance of MNP consumption and adverse event reporting (morbidity monitoring) will be done during weekly visits of the infants.

In a follow-on study, iron absorption from the two above described mentioned iron-fortified maize-based test meals will be measured in 24 infants aged 6-12 months without pre-feeding of GOS. All procedures will be done identical as described above.

ELIGIBILITY:
Inclusion Criteria:

* Age of 6-14 months at baseline
* Assessment of good health as assessed by professional staff at Msambweni District Hospital
* Willingness of their caregiver to provide informed consent

Exclusion Criteria:

* Hemoglobin <70 g/L ; these infants will be referred for treatment according to local standard of care.
* Severe underweight (Z-score weight-for-age <-3) and /or severe wasting (Z-score weight-for-height<-3)
* Chronic or acute illness or other conditions that in the opinion of the Principle Investigator (PI) or co-researchers would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Participants taking part in other studies requiring the drawing of blood
* Participants who are taking iron-containing food supplements or tablets/drops
* Participants who are taking antibiotics

Ages: 6 Months to 14 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2016-01; Primary Completion 2016-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the isotopic ratio of iron in blood at week 5 | Baseline and Week 5
  The change in the isotopic ratio of iron will be measured after the administration of test meals including iron isotopes.

SECONDARY OUTCOMES:
Gut microbiome composition | Baseline and Week 3
  The changes in the gut microbiome composition from baseline to week 3 will be compared among the two groups and correlated to the iron absorption from the test meal.
Fecal pH | Baseline and Week 3
  The changes in fecal pH from baseline to week 3 will be compared among the two groups and correlated to the iron absorption from the test meal.
Fecal short chain fatty acids (SCFAs) | Baseline and Week 3
  The changes in SCFAs from baseline to week 3 will be compared among the two groups and correlated to the iron absorption from the test meal.
H.pylori | Baseline
  H.pylori infection as determinant of iron absorption

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zimmermann, MD, Principal Investigator — Swiss Federal Institute of Technology (ETH), Zurich
Locations (1):
- Msambweni District Hopsital, Msambweni, Kwale County, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Data will be published in a peer-review journal.

REFERENCES:
- [Derived] Mikulic N, Uyoga MA, Paganini D, Mwasi E, Stoffel NU, Zeder C, Karanja S, Zimmermann MB. Consumption of a Single Dose of Prebiotic Galacto-Oligosaccharides Does Not Enhance Iron Absorption from Micronutrient Powders in Kenyan Infants: A Stable Iron Isotope Study. J Nutr. 2021 May 11;151(5):1205-1212. doi: 10.1093/jn/nxab007. PMID 33693741
- [Derived] Paganini D, Uyoga MA, Cercamondi CI, Moretti D, Mwasi E, Schwab C, Bechtler S, Mutuku FM, Galetti V, Lacroix C, Karanja S, Zimmermann MB. Consumption of galacto-oligosaccharides increases iron absorption from a micronutrient powder containing ferrous fumarate and sodium iron EDTA: a stable-isotope study in Kenyan infants. Am J Clin Nutr. 2017 Oct;106(4):1020-1031. doi: 10.3945/ajcn.116.145060. Epub 2017 Aug 16. PMID 28814396